CLINICAL TRIAL: NCT03604367
Title: Gait Mate: Examining Neural Networks Engaged During Lower Extremity Movement in the MRI
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC Center for Biomedical Research Excellence (COBRE) in Stroke Recovery (Unknown)
Responsible Party: Sponsor
Other Study IDs: 72777
Record Dates: First submitted 2018-06-28; First posted 2018-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Motor Activity
Keywords: fMRI; BOLD Signal; Rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- GAITRite assessment: Subjects will undergo the GAITRite assessment of functional walking and then complete the Functional MRI Bipedal paradigm followed by questionnaires and assessments regarding the virtual environment.
  Interventions: Device: GAITRite assessment

INTERVENTIONS:
Device: GAITRite assessment — The fMRI Bipedal Paradigm will allow investigators to study the effects treadmill-assisted gait training have on cortical control of bipedal movement in chronic stroke patients.
  Other Names: fMRI Bipedal Paradigm

SUMMARY:
Less than 50% of stroke survivors progress to independent community ambulation. Even among the stroke survivors who achieve independent ambulation, significant residual deficits persist in balance and gait speed, with 60% of persons post-stroke reporting limitations in mobility related to walking.Consequently maximizing recovery of locomotor function is the focus of neurorehabilitation efforts worldwide. A recently completed clinical trial from members of this investigative team demonstrated that 6 weeks of treadmill training elicits substantial improvements in over ground walking speed and symmetry in persons following stroke. Consistent with the goals of the South Carolina Stroke Rehabilitation Research Center (SCSRRC) and NIH Brain Initiative, the investigators now plan to investigate the effects treadmill-assisted gait training have on cortical control of bipedal movement in chronic stroke patients. Although previous investigators have assessed neural activity during simulated walking using motor imagery, motor imagery does not simulate the typical sensory feedback associated with active movement. To move the field forward, it is necessary to measure active bipedal movement in the MR-environment in healthy volunteers, before moving forward in stroke patients.

DETAILED DESCRIPTION:
The overarching goal of this Discovery Proposal is to evaluate neural activity during unipedal and bipedal movement in a cohort of healthy individuals (Aim 1).

The rigor and reproducibility will be evaluated by comparing the results of 1) active movement -Bipedal with 2) active movement -unipedal 4 and 3) imagined movement.

Dependent measures include: 1) head motion during the fMRI task, 2) BOLD signal in the ipsilateral and contralateral motor cortex during the fMRI task, 3) force applied during the fMRI task, and 4) participant feedback using a modified version of the Presence Questionnaire (a standard tool to assess ecological validity of virtual environments.

Each Aim has a development and evaluation aspect. Through this 1 year proposal the investigators will determine if the bipedal fMRI protocol (active movement) is able to engage neural networks more robustly (e.g. greater effect size) than bipedal imagery alone in Healthy Volunteers.

Specific Aim #1: Healthy volunteers: The investigators will test the hypothesis that with active bipedal movement there will be 1) no difference in head movement, but 2) greater motor cortex BOLD signal, 3) smoother force exchange between the feet, 4) higher participant satisfaction than unipedal movement or motor imagery alone. This sample size was selected based on a prior publication of imagined movement. The outcome of this aim may result in the first publication in the field to evaluate bipedal movement in an MR-environment.

ELIGIBILITY:
Inclusion criteria:

* Age 21-65
* Right hand dominant
* Able to read and understand questionnaires and informed consent

Exclusion criteria:

* Self reported history of cardiac disease, COPD or oxygen dependence, neurological and psychiatric disorders, dementia or previous stroke, major head trauma, severe visual impairment, osteoarthritis, orthopedic problems that limit passive range of motion, illegal drug or alcohol dependence, claustrophobia
* Non-mri compatible metal implants in the body
* Pregnant females

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be screened for eligibility who are right hand dominant.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
fMRI protocols will measure neural function activity during active bipedal movement in healthy volunteers | Duration of the study, approximately 1 year
  Determine if the bipedal fMRI protocol (active movement) is able to engage neural networks more robustly (e.g. greater effect size) than bipedal imagery alone in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The data from the primary outcome measurement will be shared via manuscripts and after study completion by request to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately after first publication of the results. This is estimated to be at the end of 2019.
Access Criteria: Interested parties should contact the Principal Investigator directly